CLINICAL TRIAL: NCT05115188
Title: Randomized Crossover Study Comparing the Standard Glucose Beverage and Dex4® Tablets for 2 Hour Oral Glucose Tolerance Testing in Pregnant Women With a Positive Screen on the 50g Glucose Tolerance Challenge for Gestational Diabetes
Brief Title: DIAgnosing GDM usiNg Oral Sugar InStead
Acronym: DIAGNOSIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: REB 418-2018
Record Dates: First submitted 2021-10-01; First posted 2021-11-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: It is a population-based, prospective randomized crossover study. Women who fall into the screen positive group of the 50g GCT (1 hour serum glucose of 7.8-11 mmol/L) will be offered participation in the study. 28 Participants will be recruited and will be randomly assigned using a pre-populated allocation table to take either the standard OGTT test (75g of glucose beverage) first or the alternative OGTT test (21 Dex4® tablets) first. The first test will be referred to as OGTT-1 and the second test will be referred to as OGTT-2.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-hr OGTT with glucose beverage (Other): For the 2 hour oral glucose tolerance test (OGTT), women fast for 8 hours and then consume 75g of glucose beverage, and serum glucose levels are taken at fasting, 1 and 2 hours after drinking the glucose beverage. The 75g OGTT is the gold standard and is performed for GDM diagnosis.
  Interventions: Dietary Supplement: Glucose beverage
- 2-hr OGTT with Dex4® tablets (Experimental): Participants will be asked to ingest 21 Dex4® tablets and no more than 300ml of water within 5 minutes. Blood draws will be performed at fasting (before ingesting the dextrose monohydrate tablets), as well as 1 hour after (+/- 15 minutes) and 2 hours (+/- 15 minutes) after ingesting the dextrose monohydrate tablets.
  Interventions: Dietary Supplement: Dex4/ dextrose

INTERVENTIONS:
Dietary Supplement: Dex4/ dextrose — Participants will be asked to ingest 21 Dex4® tablets and no more than 300ml of water within 5 minutes. Blood draws will be performed at fasting (before ingesting the dextrose monohydrate tablets), as well as 1 hour after (+/- 15 minutes) and 2 hours (+/- 15 minutes) after ingesting the dextrose monohydrate tablets.
  Arms: 2-hr OGTT with Dex4® tablets
Dietary Supplement: Glucose beverage — For the 2 hour oral glucose tolerance test (OGTT), women fast for 8 hours and then consume 75g of glucose beverage, and serum glucose levels are taken at fasting, 1 and 2 hours after drinking the glucose beverage. The 75g OGTT is the gold standard and is performed for GDM diagnosis.
  Arms: 2-hr OGTT with glucose beverage

SUMMARY:
The purpose of this study is to compare the positive and negative effects of Dex4® tablets, as an alternative form of fast acting carbohydrate, compared to the current standard diagnostic test, glucose beverage. The investigators hypothesis that because of their availability in solid, chewable form, variety of flavours and lack of carbonation, Dex4® tablets may result in fewer side effects than glucose beverage and provide an equivalent carbohydrate challenge for diagnosis of gestational diabetes.

DETAILED DESCRIPTION:
The project is a prospective randomized crossover study. Women who fall into the screen positive group of the 50g GCT (1 hour serum glucose of 7.8-11.0 mmol/L) will be offered participation in the study. Forty-two participants will be recruited and will be randomly assigned using a pre-populated allocation table to take either the standard OGTT test (75g of glucose beverage) first or the alternative OGTT test (21 Dex4® tablets) first. The first test will be referred to as OGTT-1 and the second test will be referred to as OGTT-2. After completing OGTT-1 at the first test appointment, a questionnaire about side effects from the first test will be completed. After completing OGTT-2 at their second test appointment, a questionnaire about side effects from the second test and test preference will be completed. Each woman will complete both tests within one week and each subject will serve as their own control. Results will be kept blinded in the case report forms until both OGTT tests are done. Serum glucose will be measured using the same internationally standardised glucose-oxidase method (RocheDiagnosis) in the Sunnybrook Biochemistry lab. After serum glucose measurement, all results will be sent to the research team but only the standard of care glucose beverage test data will appear in electronic (or classical) medical records and be used for GDM diagnosis.

The participant population consists of 28 pregnant women between 24-32 weeks' gestation who have screened positive for gestational diabetes on the 50g glucose challenge test. The main drawback to participation is that women will have to undergo two fasting, 1 hour and 2 hour glucose tests within one week. Risks involved with participating in the study include: possibility of pain, bruising, swelling or infection related to drawing blood, allergic reaction symptoms such as itching, facial swelling and anaphylaxis upon consumption if the participant has an allergy to corn based products such as dextrose. These risks will be minimized by screening patients for dextrose allergy before having them sign the informed consent form.

The benefit may not be directly to the patient as they will still need to complete the standard 75g glucose beverage test but they will be contributing to new knowledge on alternatives to the standard test that may benefit other pregnant women, including themselves, in the future.

The ultimate goal of this project is to improve women's health by 1) allowing more women to be screened for GDM and 2) providing an equivalent glucose beverage alternative with fewer side effects, making the screening process more comfortable for patients who cannot tolerate glucose beverage. Improving the tolerability of the test is important because there is growing evidence that GDM significantly increases the risk of short and long term adverse consequences for both the fetus and the mother (10,11). Accurate diagnosis may allow women to implement preventative measures such as a healthy lifestyle, which has shown to be effective in preventing T2DM in women with previous GDM (19,20). There have been recent quality control issues with the commercially available glucose beverage product (16), so this alternative test could become the standard test if the dose calibration is found to be more reliable.

Primary objective 1 (PO-1): to determine if Dex4® tablets is equivalent to glucose beverage for use in the 2-hr 75g OGTT in pregnant women between 24-32 weeks' gestation who have screened positive for GDM.

Secondary objective (SO-1): to determine if women have fewer side effects and prefer the standard (glucose beverage) OGTT test or the alternative (Dex4® tablets) OGTT test

ELIGIBILITY:
Eligibility criteria must be met by 32 weeks' gestation to allow enrollment in the study.

Inclusion Criteria:

* Positive 50g GCT result between 7.8-11.0 mmol/L
* Female
* Singleton pregnancy
* Informed consent obtained and signed

Exclusion Criteria:

* Use of steroids, terbutaline, or metformin within the last 4 weeks
* Previous diagnosis of diabetes type 1 or 2 outside of pregnancy or diagnosis with any form of diabetes prior to 20 weeks of pregnancy
* Allergy to any ingredients (including the non-medicinal ingredients) in Dex4® tablets or Glucodex solution

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Glucose values in the oral glucose tolerance test | Within 7 days
  To determine if Dex4® tablets is equivalent to glucose beverage for use in the 75g OGTT in pregnant women between 24-30 weeks gestation who have screened positive for GDM. Fasting, 1hr, and 2 hr levels from the Dex4 OGTT are within 20% of the levels from the glucose beverage OGTT.

SECONDARY OUTCOMES:
Adverse effect - nausea (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported symptoms of nausea after OGTT. Collected via questionnaire.
Adverse effect - vomiting (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported symptoms of vomiting after OGTT. Collected via questionnaire.
Adverse effect - dizziness (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported symptoms of dizziness after OGTT. Collected via questionnaire.
Adverse effect - headache (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported symptoms of headache after OGTT. Collected via questionnaire.
Adverse effect - sweating (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported symptoms of sweating after OGTT. Collected via questionnaire.
Adverse effect - other (qualitative measurement) | Within 2 hours after glucose ingestion
  Patient has self-reported other symptoms after OGTT. Collected via questionnaire.
Participant preference - qualitative measurement | Immediately after completion of both study arms
  Patient reports whether she preferred Dex4 OGTT, glucose beverage OGTT, or no preference. Collected via questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT05115188/Prot_002.pdf
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT05115188/ICF_003.pdf